CLINICAL TRIAL: NCT00049387
Title: Phase I Trial of R115777 With Radiation Therapy and Temozolomide in Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Tipifarnib, Temozolomide, and Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme or Gliosarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03106; NCI-2012-03106 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-03-C-0189; NABTC-0202; NABTC-02-02 (Other: Adult Brain Tumor Consortium); NABTC-02-02 (Other: CTEP); U01CA062399 (NIH); NCT00060879 (obsolete NCT alias)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2013-12

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — tipifarnib; Temozolomide; Radiotherapy; Radiation

ARMS (1):
- Treatment (tipifarnib, temozolomide, radiation therapy) (Experimental): See Detailed Description
  Interventions: Drug: tipifarnib; Drug: temozolomide; Radiation: radiation therapy

INTERVENTIONS:
Drug: tipifarnib — Given PO
  Other Names: R115777; Zarnestra
Drug: temozolomide — Given PO
  Other Names: SCH 52365; Temodal; Temodar; TMZ
Radiation: radiation therapy — Undergo partial brain radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation

SUMMARY:
This phase I trial is studying the side effects and best dose of tipifarnib when given together with temozolomide and radiation therapy in treating patients with newly diagnosed glioblastoma multiforme or gliosarcoma. Tipifarnib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining tipifarnib, temozolomide, and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish MTD for R115777 in combination with Temozolomide with radiation in patients not on EIAEDs.

II. To define the safety of R115777 in combination with Temozolomide with radiation in this patient population.

III. To assess for evidence of antitumor activity in this patient population.

OUTLINE: This is a multicenter, dose-escalation study of tipifarnib. Patients are stratified according to concurrent use of enzyme-inducing antiepileptic drugs (yes [closed to accrual as of 3/15/05] vs no).

COMBINATION THERAPY: Patients receive oral tipifarnib twice daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Within 5-9 days after beginning tipifarnib, patients receive oral temozolomide once daily for 6 weeks and concurrently undergo partial brain radiotherapy daily 5 days a week for 6 weeks. After completion of radiotherapy, patients proceed to adjuvant therapy.

Cohorts of 3-6 patients receive escalating doses of tipifarnib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional 10 patients are treated at the MTD.

ADJUVANT THERAPY: Patients continue to receive tipifarnib as above. With the initiation of the next planned course of tipifarnib, patients receive oral temozolomide on days 1-5. Treatment repeats every 28 days for 12 courses OR 1 year (whichever is longer) in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients with progressive disease are followed at 10 weeks and then every 4 months. Patients who complete therapy are followed every 2 months for 1 year, every 3 months for 1 year, every 4 months for 1 year, and then every 6 months thereafter until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have histologically proven intracranial Glioblastoma Multiforme (GBM) or gliosarcoma (GS)
* Diagnosis will have been established by biopsy or resection within 4 weeks prior to registration
* Patients must not have received previous radiotherapy to the brain
* Patients must not have received cytotoxic drug therapy, non-cytotoxic drug therapy, or experimental drug therapy directed against the brain tumor; patients who received Gliadel wafers will be excluded; patients may have received or be receiving corticosteroids, non-EIAEDs, analgesics, and other drugs to treat symptoms or prevent complications
* Cranial MRI or contrast CT must have been performed within 21days of study entry; the use of MRI rather than CT is preferred; the same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement; if the surgical procedure was a resection, cranial MRI or contrast CT performed with 96 hours of resection is preferred but not required; patients without measurable or assessable disease are eligible
* Patients must have a plan to begin partial brain radiotherapy within 5-9 days after beginning R115777, and within 35 days (5 weeks) of the surgical procedure that established the diagnosis; radiotherapy must be given at the Radiation Oncology Department of the registering ABTC institution; radiotherapy must be given by external beam to a partial brain field in daily fractions of 2.0 Gy, to a planned total dose to the tumor of 60.0 Gy; stereotactic radiosurgery and brachytherapy will not be allowed
* Patients must be willing to forego other drug therapy against the tumor while being treated with R115777 and temozolomide
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study; patients must sign an authorization for the release of their protected health information; patients must be registered with the Adult Brain Tumor Consortium Central Office (ABTC CO) prior to treatment with study drug
* Life expectancy > 8 weeks
* Patients must have a Karnofsky performance status of >= 60
* Patients must have adequate bone marrow function and the test must be performed within 14 days prior to registration; eligibility level for hemoglobin may be reached by transfusion
* WBC >= 3,000/µl
* ANC >= 1,500/mm^3
* Platelet count of >= 100,000/mm^3
* Hemoglobin >= 10 gm/dl
* Patients must have adequate liver function and the test must be performed within 14 days prior to registration
* SGOT < 2 times ULN
* Bilirubin < 2 times ULN
* Patients must have adequate renal function before starting therapy and the test must be performed within 14 days prior to registration
* Creatinine < 1.5 mg/dL
* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy; patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible
* This study was designed to include women and minorities, but was not designed to measure differences of intervention effects; males and females will be recruited with no preference to gender; no exclusion to this study will be based on race; minorities will actively be recruited to participate
* Patients must not have active infection
* Women must not be pregnant or Breast-feeding, and women with reproductive potential must practice adequate contraception; the anti-proliferative effects of the investigational agent may be detrimental to the developing fetus or nursing infant
* Patients must not be on chronic coumadin therapy for prior medical problems (e.g. cardiac valve prophylaxis); this is due to a presumed interaction with coumadin and ZARNESTRA leading to a significant increase in INR; patients who develop or have recently developed a deep venous thrombosis or pulmonary embolism who are on or will take coumadin will be allowed to participate; however, the investigator should be prepared to monitor patients INR closely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2002-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
MTD of tipifarnib | Week 10
  Safety variables will be summarized by descriptive statistics. Adverse events that occur will be reported for each dose level and described in terms of incidence and severity. Laboratory data will be presented by dose level at each observation time. Values outside of normal limits will be identified and their frequency calculated. Parameters will be described based on the CTCAE severity grading. Distribution by CTCAE severity grade (when applicable) and clinical relevance will be given.
Incidence of adverse events | Up to 5 years
  Safety variables will be summarized by descriptive statistics. Adverse events that occur will be reported for each dose level and described in terms of incidence and severity. Laboratory data will be presented by dose level at each observation time. Values outside of normal limits will be identified and their frequency calculated. Parameters will be described based on the CTCAE severity grading. Distribution by CTCAE severity grade (when applicable) and clinical relevance will be given.
Antitumor activity | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Cloughesy, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Adult Brain Tumor Consortium, Baltimore, Maryland, United States